CLINICAL TRIAL: NCT03528863
Title: Being Present 2.0: Web-Based Mindfulness Meditation for Gastrointestinal Cancer Patients and Caregivers
Brief Title: Web-based Mindfulness Meditation in Reducing Distress in Participants With Metastatic Gastrointestinal Cancer and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 174534; NCI-2018-00622 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-04-30; First posted 2018-05-18 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Caregiver; Metastatic Gastrointestinal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (web-based mindfulness meditation) (Experimental): Participants practice with web-based mindfulness meditation over 10-15 minute guided audio sessions for 5 days a week for 8 weeks. Participants also attend meditation webinars over 60 minutes once a week, for 8 weeks.
  Interventions: Behavioral: Online Mindfulness Meditation; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Online Mindfulness Meditation — Receive web-based mindfulness meditation
  Other Names: Online Mindful Meditation; Online Mindfulness-Based Stress Reduction (MBSR); Online Mindfulness Relaxation; Online MBSR; Web-Based Mindfulness Meditation
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well web-based mindfulness meditation works in reducing distress in both participants with gastrointestinal cancer that has spread to other parts of the body, and their caregivers. Web-based mindfulness meditation, which uses audio exercises and interactive webinars taught by trained meditation instructors, may help participants with GI cancer and their caregivers reduce distress and improve their quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and acceptability of an 8-week web-based mindfulness meditation program with live webinars among patients with a metastatic gastrointestinal (GI) cancer receiving chemotherapy and their caregivers.

SECONDARY OBJECTIVES:

I. Estimate the efficacy of an 8-week web-based mindfulness meditation program with live webinars among patients with a metastatic GI cancer receiving chemotherapy and their caregivers.

OUTLINE:

Participants practice with web-based mindfulness meditation over 10-15 minute guided audio sessions for 5 days a week for 8 weeks. Participants also attend meditation webinars over 60 minutes once a week, for 8 weeks.

After completion of study, participants are followed up at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBLE PATIENTS: Carry a diagnosis of a metastatic GI cancer
* ELIGIBLE PATIENTS: Anticipate receiving chemotherapy for at least 12 weeks total from the time of recruitment
* ELIGIBLE PATIENTS: Have an estimated life expectancy of at least 6 months, assessed by principal investigator or treating investigator
* ELIGIBLE PATIENTS: Have an Eastern Cooperative Oncology Group (ECOG) performance status between 0-2
* ELIGIBLE PATIENTS: Be able to speak and read English
* ELIGIBLE PATIENTS: Be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet (assessed by participant self-report)
* ELIGIBLE PATIENTS: Have daily access to a mobile phone capable of receiving text messages, as determined by a study investigator
* ELIGIBLE PATIENTS: Be able to provide informed consent
* ELIGIBLE CAREGIVERS: Be a spouse/partner, other family member, or a close friend of a patient who consented to participate in the Being Present 2.0 study
* ELIGIBLE CAREGIVERS: Be able to speak and read English
* ELIGIBLE CAREGIVERS: Be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet (assessed by participant self-report)
* ELIGIBLE CAREGIVERS: Have access to a mobile phone capable of receiving text messages, as determined by a study investigator
* ELIGIBLE CAREGIVERS: Be able to provide informed consent

Exclusion Criteria:

* Have a current meditation practice (> 2 episodes or > 1 hour total, weekly)
* Be currently enrolled in a stress reduction program
* Have extensive hearing loss such that ability to participate in the study would be impaired
* Have participated in the original Being Present pilot study (BP1)
* Be caregivers of patients who decline Being Present 2.0 (BP2) study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by evaluating recruitment rate | At end of enrollment (Up to 1 year)
  Number of participants approached who consent to participate
Feasibility as assessed by evaluating rate of refusal to participate | At end of enrollment (Up to 1 year)
  Number of participants refusing to consent.
Feasibility as assessed by rate of attrition | At 8 weeks post end of enrollment (Up to 1 year)
  Number of participants dropping out after start of intervention for any reason.
Acceptability as assessed by adherence to practice instructions | At 8 weeks after study start (Up to 1 year)
  Number of times participant practices during study, documented via website data capture
Acceptability as assessed by adherence to practice instructions | At 8 weeks after study start (Up to 1 year)
  Number of times participant watches recorded webinars, documented via website data capture
Acceptability as assessed by adherence to practice instructions | At 8 weeks after study start (Up to 1 year)
  Number of times patient participates in live webinars, documented via roll-call.
Acceptability as assessed by adherence to practice instructions | At 8 weeks after study start (Up to 1 year)
  Average duration of meditation session (measured in minutes), documented via website data capture.

SECONDARY OUTCOMES:
Efficacy as assessed by National Comprehensive Cancer Network (NCCN) Distress Thermometer | At baseline, week 4 and week 8 after study start (Up to 1 year)
  0 to 10, with 10 being the worst level of distress
Efficacy as assessed by National Institutes of Health Patient Reported Outcomes Measurement Information System (NIH PROMIS) | At baseline, week 4 and week 8 after study start (Up to 1 year)
Efficacy as assessed by a Five Facet Mindfulness Questionnaire Short (FFMQ-SF) | At baseline, week 4 and week 8 after study start (Up to 1 year)
Efficacy as assessed by a "Are You at Peace?" one-item spiritual probe | At baseline, week 4 and week 8 after study start (Up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Atreya, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dragomanovich HM, Dhruva A, Ekman E, Schoenbeck KL, Kubo A, Van Blarigan EL, Borno HT, Esquivel M, Chee B, Campanella M, Philip EJ, Rettger JP, Rosenthal B, Van Loon K, Venook AP, Boscardin C, Moran P, Hecht FM, Atreya CE. Being Present 2.0: Online Mindfulness-Based Program for Metastatic Gastrointestinal Cancer Patients and Caregivers. Glob Adv Health Med. 2021 Nov 3;10:21649561211044693. doi: 10.1177/21649561211044693. eCollection 2021. PMID 35174001